CLINICAL TRIAL: NCT02191215
Title: Clinical and Therapeutic Evaluation of the Infection by HIV/AIDS
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1100.1457
Record Dates: First submitted 2014-07-15; First posted 2014-07-16 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Nevirapine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Nevirapine (Viramune®)
  Interventions: Drug: Nevirapine (Viramune®)

INTERVENTIONS:
Drug: Nevirapine (Viramune®)

SUMMARY:
The aim of the Post Marketing Study (PMS) is to evaluate the efficacy and safety profile of nevirapine in the management of the HIV/AIDS in an open environment.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of HIV/AIDS, no age limits
* patients could be naïve to treatment or pretreated with other antiretroviral agents

Exclusion Criteria:

* Patients with known hypersensitivity to nevirapine or any other component of the product

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Mexican patients infected by HIV/AIDS
Sampling Method: Non-Probability Sample
Enrollment: 442 (Actual)
Dates: Start 2003-06; Primary Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
Change in body weight | Baseline, up to 90 days
Change in cluster of differentiation 4 (CD4) cell count | Baseline, up to 90 days
Change in viral load (HIV RNA) | Baseline, up to 90 days
Number of patients with adverse event | up to 90 days